CLINICAL TRIAL: NCT03005132
Title: Integrative Analysis of Human Glioblastoma Multiforme
Status: Recruiting | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Jilin University (Other); Ganzhou City People's Hospital (Other)
Responsible Party: Principal Investigator, Da Fu, Principal Investigator, Shanghai 10th People's Hospital
Other Study IDs: 2016-521-Rainy
Record Dates: First submitted 2016-12-23; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: GBM
Keywords: GBM; Integrative Analysis; WES
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Normal brain tissue: Normal brain tissue from GBM patients
  Interventions: Other: Normal brain tissue
- GBM tissues: GBM tissues from GBM patients
  Interventions: Other: Normal brain tissue
- Metastasis tissues: Metastasis tissues from GBM patients
  Interventions: Other: Normal brain tissue

INTERVENTIONS:
Other: Normal brain tissue — The investigators will extract total protein, DNA and RNA from the samples.

SUMMARY:
Integrative analysis of GBM

DETAILED DESCRIPTION:
The investigators will analyzed proteomes of paired normal brain tissues and GBM, sequenced transcriptomes, perform whole exome sequencing, and single nucleotide polymorphism (SNP) array profiling for triplets, each comprising normal brain tissue, primary GBM carcinoma, and its synchronous matched metastasis, as well as analyzed genomics of GBM characterized previously by The Cancer Genome Atlas (TCGA) to conduct integrated proteogenomic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 75 years with histologically proven GBM
* No severe major organ dysfunction
* World Health Organization (WHO) performance status of 0 or 1
* No prior cancer chemotherapy

Exclusion Criteria:

* Age ≥ 76
* Severe major organ dysfunction
* WHO performance status of >1
* Prior cancer chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with GBM
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
5 years overall survival | 5 years

SECONDARY OUTCOMES:
5 years disease-free survival | 5 years
10 years overall survival | 10 years
10 years disease-free survival | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Da Fu, PhD, Principal Investigator — Shanghai 10th People's Hospital; Xiaoming Zhong, MD, Study Director — Ganzhou City People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The investigators are willing to share data.

REFERENCES:
- [Result] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787